CLINICAL TRIAL: NCT04590703
Title: A Follow-up Study to Evaluate the Safety for the Patients With ALLO-ASC-DFU Treatment in Phase 3 Clinical Trial of ALLO-ASC-DFU-301
Brief Title: A Follow-up Study to Evaluate the Safety of ALLO-ASC-DFU in ALLO-ASC-DFU-301 Clinical Trial
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLO-ASC-DFU-303
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALLO-ASC-DFU: Subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial of ALLO-ASC-DFU-301
  Interventions: Biological: ALLO-ASC-DFU
- Vehicle sheet: Subjects with Vehicle sheet treatment in phase 3 clinical trial of ALLO-ASC-DFU-301
  Interventions: Procedure: Vehicle sheet

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to Diabetic Foot Ulcer. This study is a follow-up study without intervention.
  Groups: ALLO-ASC-DFU
Procedure: Vehicle sheet — Application of Vehicle sheet to Diabetic Foot Ulcer. This study is a follow-up study without intervention.
  Groups: Vehicle sheet

SUMMARY:
This is a follow-up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial (ALLO-ASC-DFU-301) for 24 months

DETAILED DESCRIPTION:
This is an open-label follow up study to evaluate the safety for the subjects with ALLO-ASC-DFU treatment in phase 3 clinical trial (ALLO-ASC-DFU-301) for 24 months. ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are treated with ALLO-ASC-DFU sheet or Vehicle sheet in phase 3 clinical trial of ALLO-ASC-DFU-301.
2. Subjects who are able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are considered not suitable for the study by the principal investigator.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are treated with ALLO-ASC-DFU sheet or Vehicle sheet in phase 3 clinical trial of ALLO-ASC-DFU-301.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of systemic tolerance through incidence of abnormal laboratory test results | Up to 9 months
Evaluation of incidence of clinically significant change in physical examination and vital signs | Up to 18 months
Evaluation of localized tolerance through incidence of clinically significant change about treatment area | Up to 24 months
Evaluation of incidence of adverse events | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: SeungKyu Han, MD. Ph D., Principal Investigator — Korea University Guro Hospital; KiWon Young, MD. Ph D., Principal Investigator — Nowon Eulji Medical Center, Eulji University; JunPyo Hong, MD. Ph D., Principal Investigator — Asan Medical Center; JunHyeong Kim, MD. Ph D., Principal Investigator — Keimyung University Dongsan Medical Center; Chan Kang, MD. Ph D., Principal Investigator — Chungnam National University Hospital; HyungMin Hahn, MD. Ph D., Principal Investigator — Ajou University Medical Center; ChanYeong Heo, MD. Ph D., Principal Investigator — Seoul National University Bundang Hospital; YoungKoo Lee, MD. Ph D., Principal Investigator — Soonchunhyang University Hospital
Locations (8):
- South Korea (8):
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Soonchunhyang University Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu, Gyeongsangnam-do
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul